CLINICAL TRIAL: NCT06637839
Title: A Randomized, Double-blind Study Comparing the Effects of Three Distinct High Intensity Locomotor Training Protocols on Locomotor Outcomes in Subacute Stroke Patients Undergoing Adult Inpatient Rehabilitation.
Brief Title: Optimal Dosing of High-Intensity Locomotor Training for Step Attainment and Locomotor Outcomes in Stroke Patients Undergoing Acute Inpatient Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-00889
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate-Intensity Locomotor Training Program (Experimental): Treatment will be administered for 10 consecutive 1-hour sessions over a 10-day period. Therapists will deliver the assigned intervention as part of standard care.
  Interventions: Behavioral: Moderate-Intensity Locomotor Training Program
- High-Intensity Locomotor Training Program (Experimental): Treatment will be administered for 10 consecutive 1-hour sessions over a 10-day period. Therapists will deliver the assigned intervention as part of standard care.
  Interventions: Behavioral: High-Intensity Locomotor Training Program
- High-Step Count Locomotor Training Program (Active Comparator): Treatment will be administered for 10 consecutive 1-hour sessions over a 10-day period. Therapists will deliver the assigned intervention as part of standard care.
  Interventions: Behavioral: High-Step Count Locomotor Training Program

INTERVENTIONS:
Behavioral: Moderate-Intensity Locomotor Training Program — The moderate-intensity program prescribes participants to exert 50-59% of their heart rate (HR) reserve, or a score of 13-15 on Borg's rating of perceived exertion (RPE) scale.
  Arms: Moderate-Intensity Locomotor Training Program
Behavioral: High-Intensity Locomotor Training Program — The high-intensity program prescribes participants to exert at least 60% of their heart rate (HR) reserve, or a score of 16-18 on the RPE scale.
  Arms: High-Intensity Locomotor Training Program
Behavioral: High-Step Count Locomotor Training Program — The high step count program prescribes at least 600 steps per session, at less than 50% or HR reserve, or less than 13 RPE.
  Arms: High-Step Count Locomotor Training Program

SUMMARY:
The purpose of this study is to elucidate optimal dosing for High Intensity Gait Training (HIGT) to reduce locomotor disability for those undergoing inpatient rehabilitation (IR) in the subacute phase of stroke recovery.

This is a randomized controlled trial conducted at a single IR facility. Investigators will randomize patients to receive one of two distinct HIGT interventions or a high step count intervention during standard care.

ELIGIBILITY:
Inclusion Criteria:

• Primary diagnosis of stroke

Exclusion Criteria:

* Weightbearing restrictions, uncontrolled cardiopulmonary, metabolic, infectious, or psychiatric disorders, which would preclude aerobic locomotor training
* Estimated length of stay of less than 14 days
* Non-ambulatory status prior to admission (unable to walk >50 meters)
* Pregnant

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) Score | Discharge Assessment (Day 13-14)
  The BBS is a 14-item objective assessment that static balance and fall risk in adults. Each item is rated on a scale from 0-4. The total score is the sum of responses and ranges from ranges from 0 to 56, with lower scores indicating a higher risk of falling and lower functional mobility.
Ten Meter Walk Test (10mWT) Time | Discharge Assessment (Day 13-14)
  The 10mWT is an assessment of walking speed in meters per second over a distance of 10 meters.
Six Minute Walk Test (6MWT) Distance | Discharge Assessment (Day 13-14)
  The 6MWT is a sub-maximal exercise test used to assess walking endurance and aerobic capacity. Participants walk around the perimeter of a set circuit for a total of six minutes. The measure is the total distance covered in six minutes.
Inpatient Rehabilitation Facility Patient Assessment Instrument (IRF-PAI) - Admission Quality Indicator (QI) Score: Transfers | Discharge Assessment (Day 13-14)
  The IRF-PAI QI score is an ordinal categorical variable measuring how much assistance a patient requires to complete the task (transfer) There are six categories (1-6) ranging from complete dependence of the patient on a helper to independent completion of tasks. A score of 1 is assigned to dependent patients, while a score of 6 represents independent completion of tasks by a patient.
IRF-PAI - Admission QI Score: Cumulative Ambulation | Discharge Assessment (Day 13-14)
  The IRF-PAI QI score is an ordinal categorical variable measuring how much assistance a patient requires to complete the task (ambulation) There are six categories (1-6) ranging from complete dependence of the patient on a helper to independent completion of tasks. A score of 1 is assigned to dependent patients, while a score of 6 represents independent completion of tasks by a patient.
IRF-PAI - Admission QI Score: Cumulative Stairs | Discharge Assessment (Day 13-14)
  The IRF-PAI QI score is an ordinal categorical variable measuring how much assistance a patient requires to complete the task (stairs) There are six categories (1-6) ranging from complete dependence of the patient on a helper to independent completion of tasks. A score of 1 is assigned to dependent patients, while a score of 6 represents independent completion of tasks by a patient.

SECONDARY OUTCOMES:
Number of Patients Discharged at Home | Discharge Assessment (Day 13-14)
Number of Patients Discharged at Subacute Rehabilitation Facility | Discharge Assessment (Day 13-14)
Number of Steps of Locomotor Training | Discharge Assessment (Day 13-14)
  Measurement of adherence to protocols.
Time Spent in Locomotor Training | Discharge Assessment (Day 13-14)
  Measurement of adherence to protocols.
Number of Minutes Spent in Target HR Zone | Discharge Assessment (Day 13-14)
  Measurement of adherence to protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Camillieri, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: susan.camillieri@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to susan.camillieri@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.